CLINICAL TRIAL: NCT06265402
Title: Comparison Between US Guided Retrolaminar Block and Transversus Abdominis Plane Block for Post Operative Analgesia in Patient Undergoing Abdominal Plastic Surgery
Brief Title: Retrolaminar Block Versus Tab Block in Abdomioasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hadeel Elsagheer, Elwakeel street qsm1, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Block
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrolaminar block in abdominal plastic surgery (Active Comparator): In first group induction done with general anaesthia then Patient will receive bilateral us guided rertrolaminar block then bubivacane ,25%with dexa methasone 4mg as addiditive injected on the lamina at dose 20ml injected each side
  Interventions: Procedure: Tab block versus retrolaminar block in abdominal plastic surgery
- Tab block as post operative analgesia in abdominal plastic surgery (Active Comparator): In secound group after general anaesthia induction bilateral us guided tap block with ,25%bupivacaine with dexamethasone 4mg as addiditve injected on the lamina at doses 20ml in each side
  Interventions: Procedure: Tab block versus retrolaminar block in abdominal plastic surgery

INTERVENTIONS:
Procedure: Tab block versus retrolaminar block in abdominal plastic surgery — i inject 20ml bupivacine either 4mg dead in each side

SUMMARY:
The aim of the study is to compare the analgesic efficacy of Us guided retrolaminar block versus transversus abdominis plane block in patient under going abdominal plastic surgery

DETAILED DESCRIPTION:
Pain from intra abdominal surgery is a combination of somatic and visceral pain visceral pain transmitted by autonomic nervous system via sympathetic fibers from plexuses in close proximity to the viscera them selves Regional anesthetic are commonly used to prevent or minimize these side effect the use of ultra sound nerve block are commonly use as apart of multimodal post operative analgesia The tab block is used to decrease the need of post operative analgesia in patient undergoing abdominal plastic surgery It was found an alternative approach to para vertebral block the retro laminar block is performed with us guided imaging to reduce pain post operative and need analgesia

ELIGIBILITY:
Inclusion Criteria:

- 90patients aged 18/65years of both sexes and asa physical status one two and three undergoing abdominal plastic surgery

Exclusion Criteria:

* patient refusal Patient taking analgesia of chronic illness or have history of substance abuse Patient who are unable to describe their post operative pain Patient with history of coagulabathy Un cooperative patient Patient with known allergy to study drug Patient with infection at site needle puncture Patient with decompensated hepatic renal respiratory or cardiac disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Total dose of morphine consumption in the first postoperative 24hours | First 24hours
  Total dose of morphine consumption in the first postoperative 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Hadeel Elsagheer, Principal Investigator — Tanta University
Locations (1):
- TantaU U, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No